CLINICAL TRIAL: NCT03835832
Title: Innovation of Self-Assessment Tuberculin Skin Test for Latent TB Screening in HIV Patients
Brief Title: Self-Assessment Tuberculin Skin Test
Acronym: ISAT
Status: Completed | Type: Observational
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Taksin Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: HIV-NAT 260
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Tuberculin Skin Test
Keywords: Tuberculin skin test; latent TB infection; HIV/TB co-infected participants; Sensitivity; Specificity; positive predictive value (PPV); negative predictive value (NPV)
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV-infected participants who receive TST test: 0.1 ml of tuberculin purified protein derivative will be intra-dermally inoculated on the forearm of the HIV-infected participants. They will learn how to interpret the results of the TST test. When they return to the clinic, the nurse will also interpret the results of the TST test. The results from the participants will be compared to the nurses' interpretation. We will assess the sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of the innovative method.
  Interventions: Other: The participants do not receive any intervention for this study

INTERVENTIONS:
Other: The participants do not receive any intervention for this study — The participants do not receive any intervention for this study

SUMMARY:
The research team/investigator/nurse/professional health care workers will teach the participants how to read the results for TST test. The investigator will compare the reading results done by the participants to the results read by the nurses.

DETAILED DESCRIPTION:
This is a cross-sectional study of HIV-infected patients from 2 HIV clinics in Bangkok: HIV-NAT, Thai Red Cross AIDS Research Centre and Taksin Hospital. Research team/investigator/nurse/professional health care workers will assess whether the reading of TST test between the participants and the nurses are the same or not. The investigator and team believe that the readings of the TST tests between the participants and the nurses will be the same. If the investigator and team hypothesis is correct, then this will lessen the workload of the nurses and reduce the number of times the participants have to come to the clinic to see the nurses and the doctors. This is a pilot study to test this innovative method to teach the participants to read the TST results by themselves. If this technique is successful, then the investigator and team can expand the method to other hospitals in Thailand as well as in the region.

ELIGIBILITY:
Inclusion Criteria:

1. Documented HIV-1 infection
2. Aged ≥18 years old
3. No sign and symptom of active TB

Exclusion Criteria:

1. Refuse to read TST by themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected adults with documented HIV diagnosis who do not have any signs or symptoms of active TB.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
self-assessment versus nurse reading | 6 months
  this study will assess the sensitivity of this new innovative method for reading TST
self-assessment versus nurse reading | 6 months
  this study will assess the specificity of this new innovative method for reading TST
self-assessment versus nurse reading | 6 months
  this study will assess the positive predictive value (PPV) of this new innovative method for reading TST
self-assessment versus nurse reading | 6 months
  this study will assess the negative predictive value (NPV) of this new innovative method for reading TST

SECONDARY OUTCOMES:
In house questionnaire to assess the patients' satisfaction of reading TST by themselves | 6 months
  Evaluation of patients' satisfaction in self- assessment TST by using questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Sivaporn Gatechompol, MD, Principal Investigator — HIV-NAT, Thai Red Cross - AIDS Research Centre
Locations (2):
- Thailand (2):
  - HIV-NAT, Thai Red Cross AIDS Research Centre, Bangkok
  - Taksin Hospital, Bangkok